CLINICAL TRIAL: NCT01791517
Title: Clinical and Laboratory Evaluation of Three Contact Lens Materials With Four Contact Lens Solutions
Brief Title: Clinical and Laboratory Evaluation of 3 Contact Lenses With 4 Contact Lens Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CR-5230
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2017-10

CONDITIONS: Contact Lens Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Lens A (senofilcon A) (Other): Subjects randomized to Lens A will be further randomized to 1 of 12 unique solution sequences; each subject will receive all four study solutions in a random order (Solution 1(Test), Solution 2(Test), Solution 3(Test), Solution 4(Control)).
  Interventions: Other: Solution 1 (Test); Other: Solution 2 (Test); Other: Solution 3 (Test); Other: Solution 4 (Control)
- Lens B (galyfilcon A) (Other): Subjects randomized to Lens B will be further randomized to 1 of 12 unique solution sequences; each subject will receive all four study solutions in a random order (Solution 1(Test), Solution 2(Test), Solution 3(Test), Solution 4(Control)).
  Interventions: Other: Solution 1 (Test); Other: Solution 2 (Test); Other: Solution 3 (Test); Other: Solution 4 (Control)
- Lens C (etafilcon A) (Other): Subjects randomized to Lens C will be further randomized to 1 of 12 unique solution sequences; each subject will l receive all four study solutions in a random order (Solution 1(Test), Solution 2(Test), Solution 3(Test), Solution 4(Control)).
  Interventions: Other: Solution 1 (Test); Other: Solution 2 (Test); Other: Solution 3 (Test); Other: Solution 4 (Control)

INTERVENTIONS:
Other: Solution 1 (Test) — Each subject, for each lens type (Lens A, Lens B or Lens C) will be exposed to all four lens care solution in a random order
  Other Names: Revitalens
Other: Solution 2 (Test) — Each subject, for each lens type (Lens A, Lens B or Lens C) will be exposed to each lens care solution in a random order
  Other Names: Pure Moist
Other: Solution 3 (Test) — Each subject, for each lens type (Lens A, Lens B or Lens C) will be exposed to each lens care solution in a random order
  Other Names: Biotrue
Other: Solution 4 (Control) — Each subject, for each lens type (Lens A, Lens B or Lens C) will be exposed to each lens care solution in a random order
  Other Names: Clear Care

SUMMARY:
The purpose of this study is to evaluate the clinical and laboratory performance of three brand name contact lenses with three recently introduced multipurpose lens care solutions (test solutions) as well as a peroxide disinfecting solution (control solution).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instruction set forth in this clinical protocol.
3. The subject must be between 18 and 69 years of age.
4. The subject must be willing to participate in a 9-month study.
5. The subject must require a visual correction in both eyes.
6. Subjective refraction must result in a vertex-corrected spherical contact lens prescription of +2.00D to -8.00D in each eye.
7. The subject must have best-corrected visual acuity of 0.20 or better in each eye.
8. The subject must be a current wearer of spherical soft contact lenses (no bifocal contact lenses or monovision) for at least 5 days/week and at least 8 hours/day during the month prior to enrollment.
9. The subject must require no more than -1.25D cylindrical correction in each eye after vertexing to the corneal plane.
10. The subject must have normal eye with no evidence of abnormality or disease that in the opinion of the investigator would contraindicate contact lens wear.

Exclusion Criteria:

1. Self-reported current pregnancy or lactation or plans to become pregnant during the study period (subjects who report becoming pregnant during the study will be discontinued).
2. Self-reported adverse reaction to a contact lens solution to be used in the study that in the opinion of the investigator would contraindicate use of that solution.
3. Any previous ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.).
4. Any clinically meaningful slit lamp findings contraindicating contact lens wear (e.g. equal to or greater than Grade 3 finding of edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection, blepharitis/meibomian gland dysfunction) on the study specific classification scale or any other ocular abnormality that in the opinion of the investigator would contraindicate contact lens wear.
5. Any active ocular infection.
6. Current use of topical ophthalmic medications.
7. History of binocular vision abnormality or strabismus.
8. More than occasional use of dry eye/rewetting drops (more than 2 times per day on average).
9. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV) by self-report.
10. History of severe allergic reaction or anaphylaxis.
11. Other active ocular disease that in the opinion of the investigator would contraindicate contact lens wear.
12. Employee of the investigational clinic (e.g. investigator, coordinator, technician)
13. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- University of Houston College of Optometry, Houston, Texas, United States
- University of Waterloo Centre for Contact Lens Research School of Optometry, Waterloo, Ontario, Canada
- University of Manchester, Department of Optometry & Neuroscience, Manchester, Lancashire, United Kingdom

REFERENCES:
- [Derived] Schulze MM, Srinivasan S, Hickson-Curran SB, Berntsen DA, Howarth GF, Toubouti Y, Morgan P, Nichols JJ, Jones LW; Performance of Contact Lens Solutions Study Group. Lid Wiper Epitheliopathy in Soft Contact Lens Wearers. Optom Vis Sci. 2016 Aug;93(8):943-54. doi: 10.1097/OPX.0000000000000919. PMID 27391533
- [Derived] Berntsen DA, Hickson-Curran SB, Jones LW, Mathew JH, Maldonado-Codina C, Morgan PB, Schulze MM, Nichols JJ; Performance of Contact Lens Solutions Study Group. Subjective Comfort and Physiology with Modern Contact Lens Care Products. Optom Vis Sci. 2016 Aug;93(8):809-19. doi: 10.1097/OPX.0000000000000901. PMID 27309523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 269 Subjects were enrolled into this study. Of the enrolled 33 subjects did not meet the eligibility criteria. In Phase I 28 subjects were discontinued and 208 subjects completed Phase I. Of the 208 subjects that continued into Phase II 187 subjects completed the study and 21 subjects were discontinued from the from Phase II.
Pre-assignment Details: Subjects were first randomized to 1 of 3 lenses(Lens A: senofilcon A, Lens B: galyfilcon A, Lens C: etafilcon A), then within each lens subjects were randomized to 1 of 12 unique solution sequences, totaling in 36 sequences. Due to such a large number of sequences for reporting purposes, subject disposition is reported by solution and period.
Groups:
- Biotrue/PureMoist/Revitalens/Clear Care; Biotrue/RevitaLens/Clear Care/PureMoist; Biotrue/Clear Care/PureMoist/RevitaLens; PureMoist/Biotrue/Clear Care/RevitaLens; PureMoist/RevitaLens/Biotrue/Clear Care; PureMoist/Clear Care/RevitaLens/Biotrue; RevitaLens/Biotrue/PureMoist/Clear Care; RevitaLens/PureMoist/Clear Care/Biotrue; RevitaLens/Clear Care/Biotrue/PureMoist; Clear Care/Biotrue/RevitaLens/PureMoist; Clear Care/PureMoist/Biotrue/RevitaLens; Clear Care/RevitaLens/PureMoist/Biotrue: Subjects were first randomized to receive to one of three lenses lens. For Phase I subjects were then further randomized to one of twelve unique solution sequences.
Period: Phase I: Period 1
Arm/Group | Biotrue/PureMoist/Revitalens/Clear Care | Biotrue/RevitaLens/Clear Care/PureMoist | Biotrue/Clear Care/PureMoist/RevitaLens | PureMoist/Biotrue/Clear Care/RevitaLens | PureMoist/RevitaLens/Biotrue/Clear Care | PureMoist/Clear Care/RevitaLens/Biotrue | RevitaLens/Biotrue/PureMoist/Clear Care | RevitaLens/PureMoist/Clear Care/Biotrue | RevitaLens/Clear Care/Biotrue/PureMoist | Clear Care/Biotrue/RevitaLens/PureMoist | Clear Care/PureMoist/Biotrue/RevitaLens | Clear Care/RevitaLens/PureMoist/Biotrue
Started | 19 | 20 | 20 | 19 | 20 | 20 | 20 | 20 | 20 | 20 | 18 | 20
Completed | 18 | 18 | 18 | 17 | 19 | 19 | 19 | 20 | 19 | 19 | 18 | 19
Not Completed | 1 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Lens Fitting | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Lens Handling DIfficulties | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Phase I: Period 2
Arm/Group | Biotrue/PureMoist/Revitalens/Clear Care | Biotrue/RevitaLens/Clear Care/PureMoist | Biotrue/Clear Care/PureMoist/RevitaLens | PureMoist/Biotrue/Clear Care/RevitaLens | PureMoist/RevitaLens/Biotrue/Clear Care | PureMoist/Clear Care/RevitaLens/Biotrue | RevitaLens/Biotrue/PureMoist/Clear Care | RevitaLens/PureMoist/Clear Care/Biotrue | RevitaLens/Clear Care/Biotrue/PureMoist | Clear Care/Biotrue/RevitaLens/PureMoist | Clear Care/PureMoist/Biotrue/RevitaLens | Clear Care/RevitaLens/PureMoist/Biotrue
Started | 18 | 18 | 18 | 17 | 19 | 19 | 19 | 20 | 19 | 19 | 18 | 19
Completed | 17 | 15 | 16 | 16 | 19 | 18 | 19 | 20 | 19 | 18 | 16 | 19
Not Completed | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Unsatisfactory Lens Fit | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Unsatisfactory Visual Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lens Discomfort | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I: Period 3
Arm/Group | Biotrue/PureMoist/Revitalens/Clear Care | Biotrue/RevitaLens/Clear Care/PureMoist | Biotrue/Clear Care/PureMoist/RevitaLens | PureMoist/Biotrue/Clear Care/RevitaLens | PureMoist/RevitaLens/Biotrue/Clear Care | PureMoist/Clear Care/RevitaLens/Biotrue | RevitaLens/Biotrue/PureMoist/Clear Care | RevitaLens/PureMoist/Clear Care/Biotrue | RevitaLens/Clear Care/Biotrue/PureMoist | Clear Care/Biotrue/RevitaLens/PureMoist | Clear Care/PureMoist/Biotrue/RevitaLens | Clear Care/RevitaLens/PureMoist/Biotrue
Started | 17 | 15 | 16 | 16 | 19 | 18 | 19 | 20 | 19 | 18 | 16 | 19
Completed | 17 | 14 | 16 | 15 | 18 | 18 | 19 | 20 | 19 | 18 | 16 | 18
Not Completed | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lens Discomfort | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I: Period 4
Arm/Group | Biotrue/PureMoist/Revitalens/Clear Care | Biotrue/RevitaLens/Clear Care/PureMoist | Biotrue/Clear Care/PureMoist/RevitaLens | PureMoist/Biotrue/Clear Care/RevitaLens | PureMoist/RevitaLens/Biotrue/Clear Care | PureMoist/Clear Care/RevitaLens/Biotrue | RevitaLens/Biotrue/PureMoist/Clear Care | RevitaLens/PureMoist/Clear Care/Biotrue | RevitaLens/Clear Care/Biotrue/PureMoist | Clear Care/Biotrue/RevitaLens/PureMoist | Clear Care/PureMoist/Biotrue/RevitaLens | Clear Care/RevitaLens/PureMoist/Biotrue
Started | 17 | 14 | 16 | 15 | 18 | 18 | 19 | 20 | 19 | 18 | 16 | 18
Completed | 17 | 14 | 16 | 15 | 18 | 18 | 19 | 20 | 19 | 18 | 16 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Biotrue/PureMoist/Revitalens/Clear Care | Biotrue/RevitaLens/Clear Care/PureMoist | Biotrue/Clear Care/PureMoist/RevitaLens | PureMoist/Biotrue/Clear Care/RevitaLens | PureMoist/RevitaLens/Biotrue/Clear Care | PureMoist/Clear Care/RevitaLens/Biotrue | RevitaLens/Biotrue/PureMoist/Clear Care | RevitaLens/PureMoist/Clear Care/Biotrue | RevitaLens/Clear Care/Biotrue/PureMoist | Clear Care/Biotrue/RevitaLens/PureMoist | Clear Care/PureMoist/Biotrue/RevitaLens | Clear Care/RevitaLens/PureMoist/Biotrue
Started | 17 | 14 | 16 | 15 | 18 | 18 | 19 | 20 | 19 | 18 | 16 | 18
Completed | 15 | 14 | 15 | 15 | 16 | 14 | 17 | 17 | 17 | 15 | 15 | 17
Not Completed | 2 | 0 | 1 | 0 | 2 | 4 | 2 | 3 | 2 | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Lens Handling Difficulties | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unsatisfactory Lens Fitting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pre-Existing Ocular Issue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population consists of subjects that were randomized to 1 of 3 study lenses and 1 of 12 solution sequences.
Groups:
- Etafilcon A: All subjects that were randomized to the study lens etafilcon A and 1 of 12 possible solution sequences.
- Galyfilcon A: All subjects that were randomized to the study lens galyfilcon A and 1 of 12 possible solution sequences.
- Senofilcon A: All subjects that were randomized to the study lens senofilcon A and 1 of 12 possible solution sequences.
- Total: Total of all reporting groups
Arm/Group | Etafilcon A | Galyfilcon A | Senofilcon A | Total
Number analyzed (Participants) | 80 | 78 | 78 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.33 (9.726) | 30.38 (10.091) | 29.78 (9.938) | 30.17 (9.879)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 50 | 53 | 158
  Male | 25 | 28 | 25 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18 | 18 | 22 | 58
  Black or African American | 9 | 5 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  White | 52 | 45 | 43 | 140
  Other | 1 | 10 | 6 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 28 | 26 | 26 | 80
  United States | 26 | 24 | 27 | 77
  United Kingdom | 26 | 28 | 25 | 79

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Score (Senofilcon A Lens)
Description: CLUE overall comfort is assessed using the Contact Lens User Experience (CLUE)TM questionnaire for the senofilcon A lens only. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD).
Time Frame: 2-Week Follow-up
Population: The analysis population consists of all subjects that have completed all study visits without a major protocol deviation. The number of subjects reported above is the maximum number of subjects for that solution. The number of subjects may vary per solution/lens combination, since this study was stratified by contact lens.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Solution 1(RevitaLens): Subjects that received solution 1 during any of the 4 study periods.
- Solution 2(PureMoist): Subjects that received solution 2 during any of the 4 study periods.
- Solution 3(Biotrue): Subjects that received solution 3 during any of the 4 study periods.
- Solution 4(Clear Care): Subjects that received solution 4 during any of the 4 study periods.
Arm/Group | Solution 1(RevitaLens) | Solution 2(PureMoist) | Solution 3(Biotrue) | Solution 4(Clear Care)
Number analyzed (Participants) | 69 | 69 | 69 | 69
units on a scale | 64.42 (22.536) | 59.73 (25.470) | 63.75 (21.796) | 63.47 (23.739)

2. Primary Outcome: Overall Comfort Score (Galyfilcon A Lens)
Description: CLUE overall comfort is assessed using the Contact Lens User Experience (CLUE)TM questionnaire for the galyfilcon A lens only. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD).
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solution 1(RevitaLens) | Solution 2(PureMoist) | Solution 3(Biotrue) | Solution 4(Clear Care)
Number analyzed (Participants) | 69 | 69 | 69 | 69
units on a scale | 59.79 (23.430) | 56.95 (24.679) | 58.52 (22.197) | 59.83 (22.437)

3. Primary Outcome: Overall Comfort Score (Etafilcon A Lens)
Description: CLUE overall comfort is assessed using the Contact Lens User Experience (CLUE)TM questionnaire for the etafilcon A lens only. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD).
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solution 1(RevitaLens) | Solution 2(PureMoist) | Solution 3(Biotrue) | Solution 4(Clear Care)
Number analyzed (Participants) | 65 | 65 | 65 | 65
units on a scale | 62.57 (25.158) | 67.44 (19.65) | 62.43 (21.492) | 65.33 (21.163)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 52 weeks.
Description: Adverse events from Phase I and Phase II are reported together due to the large number of lens and solution combinations.
Groups:
- Solution 1(RevitaLens): Senofilcon A: Subjects that were randomized to the senofilcon A lens and received solution 1 during any of the 4 study periods.
- Solution 1 (RevitaLens): Galyfilcon A: Subjects that were randomized to the galyfilcon A lens and received solution 1 during any of the 4 study periods.
- Solution 1(RevitaLens): Etafilcon A: Subjects that were randomized to the etafilcon A lens and received solution 1 during any of the 4 study periods.
- Solution 2(PureMoist):Senofilcon A: Subjects were randomized to the senofilcon A lens and that received solution 2 during any of the 4 study periods.
- Solution 2(PureMoist): Galyfilcon A: Subjects were randomized to the galyfilcon A lens and that received solution 2 during any of the 4 study periods.
- Solution 2(PureMoist): Etafilcon A: Subjects were randomized to the etafilcon A lens and that received solution 2 during any of the 4 study periods.
- Solution 3(Biotrue): Senofilcon A: Subjects that were randomized to the senofilcon A lens and received solution 3 during any of the 4 study periods.
- Solution 3(Biotrue): Galyfilcon A: Subjects that were randomized to the galyfilcon A lens and received solution 3 during any of the 4 study periods.
- Solution 3(Biotrue): Etafilcon A: Subjects that were randomized to the etafilcon A lens and received solution 3 during any of the 4 study periods.
- Solution 4(Clear Care): Senofilcon A: Subjects that were randomized to the senofilcon A lens and received solution 4 during any of the 4 study periods.
- Solution 4(Clear Care): Galyfilcon A: Subjects that were randomized to the galyfilcon A lens and received solution 4 during any of the 4 study periods.
- Solution 4(Clear Care): Etafilcon A: Subjects that were randomized to the etafilcon A lens and received solution 4 during any of the 4 study periods.
Arm/Group | Solution 1(RevitaLens): Senofilcon A | Solution 1 (RevitaLens): Galyfilcon A | Solution 1(RevitaLens): Etafilcon A | Solution 2(PureMoist):Senofilcon A | Solution 2(PureMoist): Galyfilcon A | Solution 2(PureMoist): Etafilcon A | Solution 3(Biotrue): Senofilcon A | Solution 3(Biotrue): Galyfilcon A | Solution 3(Biotrue): Etafilcon A | Solution 4(Clear Care): Senofilcon A | Solution 4(Clear Care): Galyfilcon A | Solution 4(Clear Care): Etafilcon A
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/78 | 0/80 | 0/78 | 0/78 | 0/80 | 1/78 | 0/78 | 1/80 | 1/78 | 0/78 | 0/80
Other Adverse Events (participants affected / at risk) | 0/78 | 0/78 | 0/80 | 0/78 | 0/78 | 0/80 | 0/78 | 0/78 | 0/80 | 0/78 | 0/78 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solution 1(RevitaLens): Senofilcon A (N=78) | Solution 1 (RevitaLens): Galyfilcon A (N=78) | Solution 1(RevitaLens): Etafilcon A (N=80) | Solution 2(PureMoist):Senofilcon A (N=78) | Solution 2(PureMoist): Galyfilcon A (N=78) | Solution 2(PureMoist): Etafilcon A (N=80) | Solution 3(Biotrue): Senofilcon A (N=78) | Solution 3(Biotrue): Galyfilcon A (N=78) | Solution 3(Biotrue): Etafilcon A (N=80) | Solution 4(Clear Care): Senofilcon A (N=78) | Solution 4(Clear Care): Galyfilcon A (N=78) | Solution 4(Clear Care): Etafilcon A (N=80)
Retro-peritoneal abscess in the kidney area. (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — According to the participant, his doctors hypothesized that the development of the abscess may be related to a perforated appendix he had in November 2011. This adverse event was deemed unrelated to the study by the investigator.
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 — Subject experienced two seizures, on August 03, 2013 to August 04, 2013. Subject has a history of seizures and stopped taking medicine(without doctor's approval). The adverse event was deemed unrelated to the study by the investigator.
Mental Health / Phychiatric Hospital Admission (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 — Subject's discontinuation of seizure medication and mental health status and was admitted to the hospital on August 03, 2013. The adverse event was deemed unrelated to the study by the investigator.
Reconstructive Surgery on Left Upper Arm (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — This event was deemed unrelated to the study by the investigator.
Viral Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Suspect viral meningitis. Had severe vomiting and headaches. Subject admitted to hospital. This was deemed unrelated to the study by the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days